CLINICAL TRIAL: NCT03106181
Title: A Randomised Controlled Trial of Cataract Surgery Versus Combined Cataract Surgery With Insertion of iStent Inject®
Brief Title: A Comparison of Cataract Surgery Alone and Cataract Surgery With iStent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Victoria Eye and Ear Hospital (Other Government)
Collaborators: Glaukos Corporation (Industry); Center for Eye Research Australia (Other)
Responsible Party: Principal Investigator, Jennifer Fan Gaskin, Ophthalmologist, Royal Victoria Eye and Ear Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: iStent RCT
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Phacoemulsification; Lens Implantation, Intraocular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cataract surgery (Active Comparator): Conventional phacoemulsification cataract surgery and intraocular lens implantation
  Interventions: Procedure: Phacoemulsification and intraocular lens implant
- Cataract surgery plus iStent inject® (Experimental): Conventional phacoemulsification cataract surgery and lens implantation plus insertion of iStent inject®
  Interventions: Device: iStent inject®; Procedure: Phacoemulsification and intraocular lens implant

INTERVENTIONS:
Device: iStent inject® — Insertion of iStent inject®
  Arms: Cataract surgery plus iStent inject®
Procedure: Phacoemulsification and intraocular lens implant — Conventional phacoemulsification cataract surgery and intraocular lens implant

SUMMARY:
This study aims to recruit patients of the Glaucoma Investigative and Research Unit (GIRU) of Royal Victorian Eye and Ear Hospital (RVEEH) with mild to moderate glaucoma who are due to undergo cataract surgery and randomise each to either cataract surgery or combined cataract surgery with iStent Inject® insertion. Only patients who meet the inclusion criteria and none of the exclusion criteria will be recruited. The outcomes measures of the study will be a comparison of: 1) extent of IOP reduction; 2) reduction in number of topical glaucoma medications; 3) patient treatment satisfaction - between the two treatment groups.

DETAILED DESCRIPTION:
Glaucoma is the commonest cause of irreversible blindness in the world. Treatment centres around lowering intraocular pressure (IOP) and typically includes medication (least invasive), laser, to surgery (most invasive). The gold-standard glaucoma operation is the trabeculectomy. Whilst it is effective at lowering IOP, it is associated with potentially devastating complications including bleb leak, hypotonous maculopathy, blebitis and endophthalmitis. In recent years, minimally- invasive glaucoma surgery (MIGS) has become an increasingly popular option of treating mild to moderate glaucoma. It is usually performed in conjunction with cataract surgery. The iStent (Glaukos Corporation, California, USA) is one of the most commonly utilised MIGS devices in the world and one of two Therapeutic Goods Administration (TGA)- approved MIGS devices in Australia. The iStent Inject® is the second generation iStent device and Australia is one of the first countries in the world to have access to this. So far there are no published randomised controlled trials comparing the effect of cataract surgery alone to combined cataract surgery with insertion of iStent Inject®.

This study aims to recruit patients of the Glaucoma Investigative and Research Unit (GIRU) of Royal Victorian Eye and Ear Hospital (RVEEH) with mild to moderate glaucoma who are due to undergo cataract surgery and randomise each to either cataract surgery or combined cataract surgery with iStent Inject® insertion. Only patients who meet the inclusion criteria and none of the exclusion criteria will be recruited. The outcomes measures of the study will be a comparison of: 1) extent of IOP reduction; 2) reduction in number of topical glaucoma medications; 3) patient treatment satisfaction - between the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Diagnosis of mild-to-moderate open angle glaucoma
* Presence of cataract requiring surgery
* Good understanding of both verbal and written English
* Able to provide informed consent

Exclusion Criteria:

* Recent intraocular surgery within last 3 months
* Other ocular pathology affecting vision
* Inability to complete the elements of the study, eg: coma, hemodynamic instability, ventilator dependence, that could be of concern in the investigator's judgment.
* Non-elective hospitalisation within the past 60 days that could be of concern in the investigator's judgment.
* Medical illness that in the judgment of the investigator would jeopardise the safe completion of the study. Examples include cancer, chronic inflammatory disease, chronic liver insufficiency, epilepsy, thrombocytosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | Up to 2 years
  Intraocular pressure reduction
Glaucoma medications | Up to 2 years
  Number of glaucoma medications

SECONDARY OUTCOMES:
Treatment satisfaction | Up to 2 years
  Patient treatment satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Fan Gaskin, FRANZCO, Principal Investigator — Royal Victoria Eye and Ear Hospital; Brian Ang, FRANZCO, Principal Investigator — Royal Victoria Eye and Ear Hospital
Locations (1):
- Royal Victorian Eye and Ear Hospital, East Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No